CLINICAL TRIAL: NCT06343701
Title: Investigation of Motor Imaging Skills in Children With Spastic Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: BAİBÜ-SAT4
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy, Spastic
Keywords: cerebral palsy; upper extremity; Imagination
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unilateral cerebral palsy: Cerebral Palsy (CP) is a group of permanent disorders in activity limitation, motor and posture development due to non-progressive damage to the developing fetus or infant brain. In spastic unilateral CP, involvement occurs unilaterally in one half of the body.
  Interventions: Other: Implicit motor imagery; Other: Explicit motor imagery
- Bilateral cerebral palsy: Cerebral Palsy (CP) is a group of permanent disorders in activity limitation, motor and posture development due to non-progressive damage to the developing fetus or infant brain. In spastic bilateral CP, involvement is seen bilaterally in all 4 extremities.
  Interventions: Other: Implicit motor imagery; Other: Explicit motor imagery
- Typically developing children: Children with typical development are children who behave in accordance with the developmental level expected for their age.
  Interventions: Other: Implicit motor imagery; Other: Explicit motor imagery

INTERVENTIONS:
Other: Implicit motor imagery — Implicit motor imagery is the ability to engage with the projection and manipulation of the body schema from a first-person perspective. Implicit motor imagery skills were evaluated Recognize App Recognize Hand Hand Laterality Task with, developed by NOI group. (http://www.noigroup.com/ Recognise).
Other: Explicit motor imagery — In explicit motor imagery, the person simulates a specific motor movement, that is, the individual is aware that she is imagining the movement.Explicit motor imagery skills were evaluated with Movement Imagery Questionnaire for Children (MIQ-C), mental chronometry and box block test.

SUMMARY:
The aim of this study was to investigate implicit and explicit motor imagery skills in children with spastic cerebral palsy and typically developing children. The main questions it aims to answer are:

* There is a difference between the implicit motor imagery skills of children with bilateral and unilateral CP.
* There is a difference between the explicit motor imagery skills of children with bilateral and unilateral CP.
* There is a difference between the implicit motor imagery skills of children with cerebral palsy and typically developing children.
* There is a difference between the explicit motor imagery skills of children with cerebral palsy and typically developing children.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a group of permanent disorders in activity limitation, motor and posture development due to non-progressive damage to the developing fetus or infant brain. Motor disorders in CP are often accompanied by sensory, perception, cognitive, communication, language and speech disorders, behavioral disorders, epilepsy, vision, hearing, endocrine, urogenital and secondary musculoskeletal system problems.

To date, CP has been classified by many researchers. The most recently used classification is the classification made by the Surveillance of Cerebral Palsy in Europe (SCPE) in 2000. According to this classification, SP; They are divided into 3 groups: spastic, dyskinetic and ataxic types. In spastic type CP, abnormal posture and movement patterns, increased muscle tone, pathological reflexes (Babinski, clonus, etc.) are dominant. The most common type of CP is spastic type CP. Spastic type CP is divided into bilateral and unilateral CP. Involvement in spastic bilateral CP, bilaterally in 4 extremities; In spastic unilateral CP, involvement occurs unilaterally in one half of the body. Dyskinetic type SP; It is characterized by abnormal posture and movement patterns, involuntary, uncontrollable, often stereotypic movements. It is divided into two groups: dystonic and choreoathetoid CP. While hypokinesia and hypertonus predominate in dystonic type CP, hyperkinesia and hypotonus predominate in choreoathetoid type CP. Ataxic type CP is characterized by coordination disorder in target-directed movements, gait and trunk control deficiencies, intention tremor, and speech disorder.

Recent studies indicate that motor disorders in children with CP are not only related to movement execution, but also to impairments in cognitive process, motor planning including motor control, and motor imagery ability.

Motor imagery refers to a mental process in which the individual mentally imagines a movement without actually performing an active movement. Studies have shown that similar brain regions are activated during movement performance and movement visualization. Motor imagined movements and actively performed motor movements occur in the premotor and parietal areas, basal ganglia and cerebellum. Based on this, motor imagery allows identifying the cognitive and cerebral properties of movement representation independently of motor output and sensory feedback.

Imagination is divided into two: express and implicit motor imagery. During express motor imagery, the person simulates a specific motor movement, that is, the individual is aware that he is visualizing the movement. Implicit motor imagery is the ability to engage with the projection and manipulation of the body schema from a first-person perspective. In implicit motor imagery, the movement is visualized unconsciously.

Implicit motor imagery skills will be evaluated Hand Laterality Task, Explicit motor imagery skills will be evaluated with Movement Imagery Questionnaire for Children (MIQ-C), mental chronometry and box block test. All assessments will be evaluated and recorded separately in the dominant and nondominant upper extremities as actual performance and imaged performance.

All evaluations will be made in between the ages of 6-18 typically developing children and children with unilateral and bilateral cerebral palsy with level 1 or 2 according to the Gross Motor Function Classification System (GMFCS), Manual Ability Classification System (MACS), Communication Function Classification System (CFCS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spastic type CP between the ages of 6-18
* Gross Motor Function Classification System (GMFSS) level 1- 2
* Manual Dexterity Classification System (EBSS) level 1-2
* Having at least 24 points from the Mini-Mental test for children,
* Having an IQ > 70,
* To be able to understand the instructions of the study.

Exclusion Criteria:

* Having severe vision, hearing or attention problems,
* Having advanced cardiovascular or cognitive problems,
* Not being able to follow work instructions,
* Having had upper extremity surgery within the last 6 months,
* Having received MI training in the last 6 months.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study included between the ages 6 and 18 years 10 children with unilateral and bilateral cerebral palsy with level 1 or 2 according to the Gross Motor Function Classification System (GMFCS), Manual Ability Classification System (MACS), Communication Function Classification System (CFCS) and 10 typically developing children.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-05-05 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
Explicit motor imagery -1 | two years
  Box and block test,Participants were first asked to pass the maximum number of wooden blocks to the other side of the wooden box in 60 seconds, three times for each hand. The actual number of movement blocks was obtained by calculating the average of 3 applications. Then, each participant was asked to visually pass the maximum number of wooden blocks to the other side of the wooden box without moving, three times for both hands. While visualizing, the participants pressed the button in front of them for each wooden block they placed, thus the number of wooden blocks they imagined passing to the other side was seen. The number of imaged movement blocks was obtained by taking the average of 3 applications. The number of wooden blocks passed with actual movement and imagined movement was compared.

SECONDARY OUTCOMES:
Explicit motor imagery - 2 | two years
  Box and block test, mental chronometry, The mental chronometry paradigm was evaluated using the wooden box and 10 wooden blocks of the box block test. The participants were first asked to grasp 10 wooden blocks from one side of the wooden box and pass them to the other side, three times in both hands, and the time taken was calculated with a stopwatch. Then, they were asked to visualize passing 10 wooden blocks to the other side of the wooden box, 3 times for each hand, and to say when they imagined that all 10 wooden blocks had passed. When they said they were done, the stopwatch was stopped. The application was performed three times on the dominant and non-dominant sides for real and imagined movements, and the average was noted. Delta time was calculated based on real and imagined movement time. . Delta time is calculated with the formula =[(real movement-imagined movement) / [(real movement+imagined movement) / 2]x100.
Explicit motor imagery - 3 | two years
  Movement Imagery Questionnaire for Children (MIQ-C),The Movement Imagination Questionnaire for Children will be used to measure visual (intrinsic, extrinsic) and kinesthetic imagery ability. It contains a total of 12 items: 4 items on internal, 4 items on external, and 4 items on kinesthetic visualization skills. Within the scope of the survey, the individual will be asked to visualize 4 different movements from 3 different visualization perspectives. The individual will be expected to first actually perform the movement in the instruction once and then imagine doing the movement. The clarity of this imagery will be rated using a Likert-type scale from 1 (very difficult to feel) to 7 (very easy to feel). A higher score from the test indicates higher imagination ability.
Implicit motor imagery | two years
  Hand Laterality Task, Implicit motor imagery capacity was assessed with the Laterality Task (choice task). Laterality task is based on deciding which side of the photograph belongs to the limb shown. Recognize Hand is an application developed by the NOI group and used to evaluate right-left discrimination.(http://www.noigroup.com/ Recognise). In terms of imagination ability and hand laterality, the sharpness of the choices made in right-left discrimination (percentage of correct answers) and the reaction time during the choice were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Ayaz Taş, Phd, Principal Investigator — Abant Izzet Baysal University
Locations (3):
- Turkey (Türkiye) (3):
  - Kdz. Ereğli Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Zonguldak, Ereğli
  - Bolu Abant İzzet Baysal University, Bolu, Gölköy/ Bolu
  - Düzce Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Düzce, Merkez

IPD SHARING:
Plan to Share IPD: No